CLINICAL TRIAL: NCT01198093
Title: Clinical Research Center for Dementia of South Korea (CREDOS)
Brief Title: Clinical Research Center for Dementia of South Korea (CREDOS)(or CRCD)
Acronym: CREDOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Principal Investigator, Doh Kwan Kim, Professor, Samsung Medical Center
Other Study IDs: 2005-02-008
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-09

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; Mild Cognitive Impairment; cohort study
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma and DNAs were prepared
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objective of this study is to present evidence-based medicine for development of clinical practice guideline through prospective study of Alzheimer's disease(AD) and mild cognitive impairment(MCI) in korea

DETAILED DESCRIPTION:
The specific aims of this study is (1) construction & maintenance of cohort for Alzheimer's disease(AD) and mild cognitive impairment(MCI); (2) study of epidemiology, rate of progression, risk factor, prognostic factor; (3) study of biomarker such as neuropsychological assessment, peripheral & CSF markers, neuroimaging(both structural & functional)

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's disease(AD) and mild cognitive impairment(MCI)will be enrolled in the study.

  1. the diagnostic criteria of Alzheimer's disease(AD) according to DSM IV or NINCDS -ADRDA
  2. the diagnostic criteria of mild cognitive impairment(MCI) A. Memory or other cognitive complaint preferably corroborated by an informant B. Objective memory impairment or other cognitive for age and education C. Largely intact general cognitive function D. Essentially preserved ADL E. Not demented

Exclusion Criteria:

* Exclusion criteria are current neurological or other psychiatric disorders, as well as a history of epileptic seizures, substantial brain damage or neurosurgical operation, according to established safety criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. Patient populatin who is suffering from memory impairment
  2. Normal subjects matched with age and gender
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2005-11; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Doh K KIm, Ph.D, Principal Investigator — Ministry of Health and Welfare
Locations (1):
- Samsung Medical Center, Seoul, Kangnam-Ku, South Korea

REFERENCES:
- [Derived] Lee YM, Park JM, Lee BD, Moon E, Jeong HJ, Chung YI, Kim JH, Kim HJ, Mun CW, Kim TH, Kim YH. Gray matter volumes and treatment response of psychotic symptoms to risperidone in antipsychotic-naive Alzheimer's disease patients. J Clin Psychiatry. 2016 Jan;77(1):e8-13. doi: 10.4088/JCP.14m09740. PMID 26845282
- [Derived] Yoon B, Shim YS, Cheong HK, Hong YJ, Lee KS, Park KH, Ahn KJ, Kim DJ, Kim YD, Choi SH, Yang DW. White matter hyperintensities in mild cognitive impairment: clinical impact of location and interaction with lacunes and medial temporal atrophy. J Stroke Cerebrovasc Dis. 2014 May-Jun;23(5):e365-72. doi: 10.1016/j.jstrokecerebrovasdis.2013.12.040. Epub 2014 Feb 28. PMID 24589036